CLINICAL TRIAL: NCT04769232
Title: Endoscopic Characterisation of Inflammatory Activity in EoE: Comparison of Two Gastroscopes With High Magnification to the Goldstandard Histology
Brief Title: Endoscopic Characterisation of Inflammation in EoE
Acronym: ECI-EoE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2020-00817
Record Dates: First submitted 2021-01-29; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Imaging (Active Comparator): In 20 randomly assigned patients, the area of endoscopically highest activity will be biopsied as determined by standard imaging. A total of 10 biopsies will be taken in 4 sets: 1 = one single biopsy at best guess of highest activity; 2 = one single biopsy at second best guess of highest activitiy, 3 = 4 biopsies in proximal esophagus with presumed activity, 4 = 4 biopsies in distal esophagus with presumed activity. Overall qualitative (eosinophilic inflammation present vs. absent) and semi-quantitative (estimation of the number of eosinophilic neutrophils according to the following categories 1: 0, 2: 1-6, 3. 7-14, 4. 15-50, 5. :50-100, 6. > 100, together with an estimation of an absolute number of eosinophilic neutrophils) inflammatory activity will be rated for the presumed localization of maximal histologic activity and subsequently for all other 10 biopsies using this imaging modality by endoscopist.
  Interventions: Device: EG-760Z endoscope by Fujifilm
- High Magnification Imaging (Experimental): In 20 randomly assigned patients, the area of endoscopically highest activity will be biopsied as determined by high magnification imaging. A total of 10 biopsies will be taken in 4 sets: 1 = one single biopsy at best guess of highest activity; 2 = one single biopsy at second best guess of highest activitiy, 3 = 4 biopsies in proximal esophagus with presumed activity, 4 = 4 biopsies in distal esophagus with presumed activity. Overall qualitative (eosinophilic inflammation present vs. absent) and semi-quantitative (see above) inflammatory activity will be rated for the presumed localization of maximal histologic activity and subsequently all other 10 biopsies using this imaging modality by endoscopist.
  Interventions: Device: EG-760Z endoscope by Fujifilm

INTERVENTIONS:
Device: EG-760Z endoscope by Fujifilm — Within a single endoscopic procedure under propofol sedation, images of the esophageal wall will be acquired and biopsies will be taken. All patients will be examined using the EG-760Z endoscope by Fujifilm.
  In all patients as part of the clinical routine 4 biopsies of the proximal and 4 biopsies of the distal esophagus will be taken.

SUMMARY:
In this study, we plan to investigate the accuracy of the EG-760Z endoscope (135x zoom) compared with standard imaging with histology as gold standard in detecting and grading inflammatory activity in patients with eosinophilic esophagitis (EoE).

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EoE) is a chronic-inflammatory disease of the esophagus. If left untreated, eosinophilic inflammation induces fibrosis, angiogenesis and stricture formation, finally resulting in a so called remodelling with structural and functional damage of the organ. In addition, patients with untreated EoE are permanently at risk of experiencing food impactions. It is therefore widely accepted that active EoE should be recognized and treated as such. Any treatment applied in EoE should ideally achieve two therapeutic goals: first, resolution of symptoms, and, second, control of inflammation.

However, in some cases of EoE, there is a dissociation between symptoms and histological response.

Furthermore, characteristic endoscopic findings may occur together but are not all seen in every EoE patient. As an example, in 7% to 10% of cases the esophagus may appear normal. Lastly, inflammatory infiltration of the esophageal wall may be discontinuous. In order to define endoscopic activity of EoE in a standardized fashion, the endoscopic reference score (EREFS) is usually applied.

Several endoscopic ﬁndings, including linear furrows, concentric rings, white exudates, decreased vasculature in the esophageal mucosa, esophageal strictures, and the esophagus of narrow caliber have been reported to be the characteristic ﬁndings of EoE, although neither of these is speciﬁc. According to a meta-analysis from 2012, consisting primarily of retrospective studies involving adult cohorts, the overall pooled prevalence of endoscopic ﬁndings in patients with EoE was 44% rings, 21% strictures, 9% narrow caliber esophagus, 48% linear furrows, 27% white exudates, and 41% decreased vascularity, with a wide variation in the prevalence of those endoscopic ﬁndings between each report.

Lastly, inflammatory infiltration of the esophageal wall may be discontinuous. Taken together, endoscopic recognition of EoE remains a major clinical challenge and diagnosis still relies on histological sampling which in turn renders the diagnosis prone to sampling errors.

In addition to that, it is well known that optimal control of inflammatory activity is crucial in order to prevent progression of fibrosis. Therefore, monitoring inflammatory activity (determined by the EoE histologic scoring system; EoE-HSS) is part of clinical routine in patients with EoE. As outlined above, endoscopic assessment, however, does not reliably reflect the underlying process of the disease during the index endoscopy and cannot be regarded as reliable follow-up test.

The investigators hypothesize that novel endoscopic technologies overcome the shortcomings of the standard endoscopic imaging. It is therefore planned to compare images of the esophageal mucosa using the EG-760Z endoscope by Fujifilm (Fujifilm Europe, Düsseldorf, Germany) to standard imaging with high magnification imaging. This novel endoscope acquires images with a magnification by a factor of 135. As gold standard, histological assessment of the inflammatory activity will be used.

ELIGIBILITY:
Inclusion Criteria:

Eligible are patients with histology-proven EoE in whom a follow-up endoscopy is indicated. Indications for follow-up endoscopy are i) determination of the response to PPI-Trial or ii) inadequate symptomatic relief despite established therapy.

Type of treatment, or response to, have no implications on eligibility.

Participants fulfilling all of the following inclusion criteria are eligible for the study:

* Patient is capable of giving informed consent
* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Have histology proven EoE and are due to undergo follow-up gastroscopy or are due to undergo gastroscopy to investigate dyspepsia (control group)
* Male and Female patients 18 years to 80 years of age

Exclusion Criteria:

* Contraindications to outpatient gastroscopy
* Contraindication for Non-anesthesia Provider Procedural Sedation and Analgesia: ASA class III or higher, morbid obesity (BMI > 40 kg/m^2), severe OSAS
* Contraindications to tissue sampling: oral anticoagulation in combination with antiaggregant such as aspirin or clopidogrel,
* Patients without subcutaneous veins that allow for insertion of peripheral venous catheters
* Women who are pregnant or breast feeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Participation in another study with investigational drug/device within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
High magnification leeds to more accurate histologic sampling | 6 months
  High magnification by a factor of 135, using the EG-760Z endoscope by Fujifilm, enables biopsies in areas with higher degree of inflammation.
  Biopsies will be analyzed by an experienced pathologist in the field of EoE. The pathologist will count the number of eosinophilic neurtophils in a high-power field (HPF). The absolut number of eosinophilic neutrophils per HPF will be compared to biopsies taken with standard imaging.

SECONDARY OUTCOMES:
Target biopsies are non-inferior to standard biopsies | 6 months
  Target single biopsies with high magnification by a factor of 135, using the EG-760Z endoscope by Fujifilm, in the proximal and distal esophagus are non-inferior to goldstandard biopsies taken with a standard endoscope (4 biopsies proximally and distally) in disease monitoring.
  Biopsies will be analyzed by an experienced pathologist in the field of EoE. The pathologist will count the number of eosinophilic neurtophils in a high-power field (HPF). The absolut number of eosinophilic neutrophils per HPF will be compared to biopsies taken with standard imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Biedermann, Principal Investigator — Universitätsspital Zürich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Straumann A. Medical therapy in eosinophilic oesophagitis. Best Pract Res Clin Gastroenterol. 2015 Oct;29(5):805-814. doi: 10.1016/j.bpg.2015.06.012. Epub 2015 Jul 26. PMID 26552779
- [Background] Bisschops R, Hassan C, Bhandari P, Coron E, Neumann H, Pech O, Correale L, Repici A. BASIC (BLI Adenoma Serrated International Classification) classification for colorectal polyp characterization with blue light imaging. Endoscopy. 2018 Mar;50(3):211-220. doi: 10.1055/s-0043-121570. Epub 2017 Oct 24. PMID 29065437
- [Background] Kim HP, Vance RB, Shaheen NJ, Dellon ES. The prevalence and diagnostic utility of endoscopic features of eosinophilic esophagitis: a meta-analysis. Clin Gastroenterol Hepatol. 2012 Sep;10(9):988-96.e5. doi: 10.1016/j.cgh.2012.04.019. Epub 2012 May 18. PMID 22610003
- See also: Clinical investigation of medical devices for human subjects -- Good clinical practice — https://www.iso.org/home.html